CLINICAL TRIAL: NCT03828695
Title: Efficacy and Efficiency of Uterocervical Angle for Prediction of Preterm Labor in Patients With Idiopathic Polyhydramnios: a Prospective Cohort Study
Brief Title: Uterocervical Angle in Idiopathic Polyhydramnios
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nefise Nazlı YENIGUL (Other)
Responsible Party: Sponsor-Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecology, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Organization: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 10988
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- uterocervical angle (Other): uterocervical angle is the angle between lower segment of uterus and cervix
  Interventions: Other: uterocervical angle

INTERVENTIONS:
Other: uterocervical angle — uterocervical angle is the angle between lower segment of uterus and cervix

SUMMARY:
To evaluate the performance of uterocervical angle (UCA) in the prediction of preterm labor in isolated polyhydramnios

ELIGIBILITY:
Inclusion Criteria:

* isolated polyhydramnios pregnancies
* no previous systemic illnesses

Exclusion Criteria:

* abnormal Pap smear
* previous cesarean section
* history of dilatation and curettage (D&C)
* history of loop electrosurgical excision procedure (LEEP) and cervical conization

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
prediction of preterm birth by uterocervical angle in patients with idiopathic polyhydramnios. | 6 month
  During the study period, women were enrolled and uterocervical angle were measured in the first evaluations of polyhydramnios patients in policlinics. Routine pregnancy follow-up was done by our team and weeks of delivery and maternal-fetal outcomes were noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise N YENIGUL, Sanliurfa, Turkey (Türkiye)